CLINICAL TRIAL: NCT01526941
Title: A Double-blind, Randomised, Two-Period Crossover Trial Comparing the Single Dose and Steady State Pharmacodynamics of Biphasic Insulin Aspart 30 and Biphasic Insulin Aspart 70 in Subjects With Type 1 Diabetes
Brief Title: Comparison of Single Dose and Steady State Pharmacodynamics of Biphasic Insulin Aspart 30 and 70 in Subjects With Type 1 Diabetes
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: BIASP-1318
Record Dates: First submitted 2012-02-01; First posted 2012-02-06 (Estimated); Last update posted 2017-01-05 (Estimated); Status verified 2017-01

CONDITIONS: Diabetes; Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 1 | interventions — insulin aspart, insulin aspart protamine drug combination 30:70

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment period 1 (Experimental)
  Interventions: Drug: biphasic insulin aspart 30; Drug: biphasic insulin aspart 70
- Treatment period 2 (Experimental)
  Interventions: Drug: biphasic insulin aspart 30; Drug: biphasic insulin aspart 70

INTERVENTIONS:
Drug: biphasic insulin aspart 30 — Dose individually adjusted. Administered subcutaneously (s.c., under the skin) three times a day for 1 week in each treatment period. A wash-out period of 2-6 weeks will take place between treatment periods
Drug: biphasic insulin aspart 70 — Dose individually adjusted. Administered subcutaneously (s.c., under the skin) three times a day for 1 week in each treatment period. A wash-out period of 2-6 weeks will take place between treatment periods

SUMMARY:
This trial is conducted in Europe. The aim of this trial is to compare the single dose and steady state pharmacodynamics of biphasic insulin aspart 30 and biphasic insulin aspart 70 in subjects with type 1 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 diabetes for at least 12 months
* Currently on basal bolus treatment with soluble human insulin, Lispro and NPH insulin or Lantus. NPH insulin may be administered once or twice daily
* BMI (Body Mass Index) maximum 35 kg/m^2
* Able and willing to perform self-blood glucose monitoring

Exclusion Criteria:

* The receipt of any investigational drug within the last 30 days prior to this trial
* Total daily insulin dose at least 1.8 U/kg/day
* Currently being treated with insulin aspart products
* A history of drug abuse or alcohol dependence within the last 5 years
* Impaired hepatic function
* Impaired renal function
* Blood donation (exceeding 500 ml) within the last nine weeks or haemoglobin below the lower reference limit according to the local laboratory
* Cardiac problems
* Severe, uncontrolled hypertension

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2001-05; Primary Completion 2001-07 (Actual); Study Completion 2001-07 (Actual)

PRIMARY OUTCOMES:
Steady state area under the glucose infusion rate profile, 6-12 hours

SECONDARY OUTCOMES:
GIRmax, the maximal glucose infusion rate value
tmax, time to maximum glucose infusion rate value
area under the glucose infusion rate profile
Time to 50% of area under the glucose infusion rate profile, 0-12 hours
Cmax, maximum concentration
tmax, time to reach Cmax
Area under the curve
t½, terminal half-life
Adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR,1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Neuss, Germany

REFERENCES:
- [Result] Bott S, Tusek C, Heinemann L, Friberg HH, Heise T. The pharmacokinetic and pharmacodynamic properties of biphasic insulin Aspart 70 (BIAsp 70) are significantly different from those of biphasic insulin Aspart 30 (BIAsp 30). Exp Clin Endocrinol Diabetes. 2005 Oct;113(9):545-50. doi: 10.1055/s-2005-872852. PMID 16235159
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com